CLINICAL TRIAL: NCT05738993
Title: A Double-Blind, Comparative, Randomized Clinical Study of the Pharmacokinetics, Safety, and Immunogenicity of a Single Intravenous Infusion of BCD-178 or Perjeta® in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-178-1
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-178 group (Experimental): single IV infusion of BCD-178 at a dose of 420 mg
  Interventions: Drug: BCD-178
- Perjeta Group (Active Comparator): single IV infusion of Perjeta at a dose of 420 mg
  Interventions: Drug: Perjeta

INTERVENTIONS:
Drug: BCD-178 — A single intravenous (IV) infusion at a dose of 420 mg
  Other Names: pertuzumab
  Arms: BCD-178 group
Drug: Perjeta — A single intravenous (IV) infusion at a dose of 420 mg
  Other Names: pertuzumab
  Arms: Perjeta Group

SUMMARY:
This is a double-blind, comparative, randomized phase I study comparing pharmacokinetics, safety and immunogenicity profiles of a biosimilar pertuzumab (BCD-178) and Perjeta after a single intravenous infusion in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Men aged 18-45 years;
* Body mass index (BMI) in the range of 18.5 30.0 kg/m2;
* The confirmed "healthy" status;
* Left ventricular ejection fraction (LVEF) > 50 % based on the results of EchoCG at screening;
* Willingness of the volunteers and their sexual partners of childbearing potential to use reliable methods of contraception, starting from signing the informed consent form, during the study, and for 6 months after the drug administration;

Exclusion Criteria:

* Known allergy or intolerance to monoclonal antibody products (murine, chimeric, humanized, fully human) or any other components of the study drugs;
* Values of standard laboratory and instrumental parameters exceeding the normal limits accepted at the study site;
* History or evidence of any chronic disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
AUC0-∞ | pre-dose to day 91, 23 timepoints
  Area under the concentration-time curve of the drug over the time interval from zero to infinity

SECONDARY OUTCOMES:
Cmax | pre-dose to day 91, 23 timepoints
  maximum observed plasma concentration of the drug
Tmax | pre-dose to day 91, 23 timepoints
  time from administration to maximum observed plasma concentration of the drug
T½ | pre-dose to day 91, 23 timepoints
  Elimination half-life
Kel | pre-dose to day 91, 23 timepoints
  elimination rate constant
CL | pre-dose to day 91, 23 timepoints
  total clearance
Vd | pre-dose to day 91, 23 timepoints
  volume of distribution
safety assessment | Day 1 to day 91
  frequency, severity, and profile of adverse events
immunogenicity assessment | pre-dose to day 91, 5 timepoints
  binding anti-drug antibodies (BAb) and neutralizing anti-drug antibodies (NAb)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - City Polyclinic №77, Saint Petersburg
  - X7 Clinical Research, Saint Petersburg